CLINICAL TRIAL: NCT02961894
Title: Revolution™ Peripheral Atherectomy System for Lower Extremity Peripheral Arterial Revascularization
Acronym: REVEAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rex Medical (Industry)
Collaborators: Syntactx (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REX-US-2017-001
Record Dates: First submitted 2016-11-07; First posted 2016-11-11 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Peripheral Artery Disease
Keywords: Atherectomy; Atherosclerosis
MeSH Terms: conditions — Peripheral Arterial Disease; Atherosclerosis | interventions — Atherectomy; Atherectomy, Coronary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Revolution Treatment Arm (Experimental): This is a single-arm study. All eligible and participating patients will be treated wit the Revolution™ Peripheral Atherectomy System.
  Interventions: Device: Revolution™ Peripheral Atherectomy System

INTERVENTIONS:
Device: Revolution™ Peripheral Atherectomy System — The Rex Medical Revolution™ Peripheral Atherectomy System is a minimally invasive catheter-based atherectomy system used to treat patients who suffer from PAD. This system is designed to treat a broad range of plaque types both above and below the knee and may address many of the limitations associated with existing treatment options.
  Other Names: Revolution Peripheral Atherectomy System; Percutaneous Transluminal Atherectomy; Rotational Atherectomy

SUMMARY:
To evaluate the safety and effectiveness of the Revolution™ Peripheral Atherectomy System in the treatment of infrainguinal lower extremity peripheral arterial occlusive disease.

This Atherectomy system will be used on eligible patients with stenosis of at least 70% diameter reduction to evaluate the change in stenosis after the procedure (effectiveness) and the presence of any major adverse events (safety) for up to 30 days after the procedure.

DETAILED DESCRIPTION:
This study intends to enroll up to 121 subjects at up to 18 investigational sites in the United States. This is a single-arm study of the Revolution™ Peripheral Atherectomy System in subjects with peripheral arterial disease (PAD).

The primary safety endpoint is freedom from 30-day Major Adverse Events (MAE), defined as the composite of all-cause mortality, clinically-driven target lesion revascularization (TLR), major target limb amputation, major target vessel perforation requiring surgical or endovascular repair and clinically-significant distal embolization in the target limb; as adjudicated by the independent Clinical Events Committee (CEC).

The primary effectiveness endpoint is technical success, defined by ≤50% diameter stenosis after atherectomy with the Revolution™ Peripheral Atherectomy System and prior to adjunctive therapy, as measured by the independent core laboratory on the post-atherectomy contrast angiogram. Effectiveness will be assessed for investigator-identified target lesions and will be calculated as a binary variable as the proportion of target lesions with technical success.

The following will be assessed as secondary endpoints of the study:

1. Change in % stenosis after treatment with Revolution™ Peripheral Atherectomy System, determined after atherectomy and prior to other adjunctive therapies, as measured by the angiographic core laboratory.
2. Procedural success as defined by target lesion residual stenosis of <30% at the conclusion of the index procedure, after atherectomy and any adjunctive endovascular treatment, as measured by the angiographic core laboratory.
3. Assessment of the individual components of the primary safety endpoint (MAE); including all-cause mortality, major target limb amputation, clinically significant distal embolization, major target vessel perforation requiring surgical or endovascular repair, and clinically-driven TLR, measured through 30 days and at 6 months.
4. Minor unplanned target limb amputation rate through 30 days and 6 months;
5. Myocardial infarction through 30 days and 6 months;
6. Incidence of target vessel revascularization (TVR) through 30 days and 6 months;
7. Frequency of angiographic procedural distal embolization (symptomatic) in the target limb as confirmed angiographically by the core laboratory;
8. Primary patency of the target lesion at 30 days and 6 months, determined by duplex ultrasound or angiography;
9. Primary-assisted patency of the target lesion at 30 days and 6 months, determined by duplex ultrasound or angiography;
10. Secondary patency of the target lesion at 30 days and 6 months, determined by duplex ultrasound or angiography.

Subjects with symptomatic PAD eligible for treatment with the Revolution™ Peripheral Atherectomy System with atherosclerotic lesions of the superficial femoral, popliteal and tibial arteries will be eligible for inclusion in the study.

A performance goal of 80% for safety and 76% for effectiveness has been established from prior studies. Enrollment of 121 subjects will provide 90% power, based upon a one-sided 97.5% exact binomial test, an anticipated 30-day MAE rate of 9%, acute technical success of 86%, and a 30-day attrition rate of approximately 10%.

The regulatory submission will be based on an approximate sample size of 121 subjects. Assuming a lesion-to-subject ratio of 1.5, approximately 165 target lesions will be evaluable for the primary effectiveness endpoint. Subset analyses will be performed for device effectiveness for superficial femoral/popliteal and tibial artery target lesions.

Pre-Enrollment procedures include testing, reviewing Medical history, physical examination with vital signs and directed peripheral vascular examination, laboratory assessment, ankle-brachial or toe-brachial index, and patient-reported outcome measures. The diagnostic angiogram at time of the planned index procedure is performed prior to the point of enrollment in the study; eligibility is, in part, based upon the anatomic findings of the angiogram.

Subjects will have required follow-up evaluations at the following time points:

1. Discharge;
2. 1 month post index procedure;
3. 6 months post index procedure;

Follow-Up Data Collection:

1. Adverse Events at the index procedure, hospital discharge, and through 6 months;
2. Rutherford Classification at 1 and 6 months;
3. Ankle-brachial or toe-brachial index at 1 and 6 months;
4. Duplex ultrasound of the target vessel at 1 and 6 months.

An independent Clinical Events Committee (CEC) will review all primary safety endpoint events, unanticipated adverse device effects, and other important safety occurrences as specified in the CEC Charter. Additionally, an independent Data Safety Monitoring Board (DSMB) will review safety data from the study at predetermined time points and as deemed necessary by the Sponsor or the DSMB Chair. The DSMB will make recommendations on protocol modifications and continuation of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Willing and able to provide informed consent.
3. Ability to take at least one form of anti-platelet therapy.
4. Rutherford categories 2 to 5 in the target limb.
5. Lesions to be treated with the study device must be located in the same limb.
6. Target lesion(s) located within the superficial femoral, popliteal or tibial arteries.
7. Target lesion(s) with stenosis ≥70% diameter reduction as measured by site-reported angiography.
8. Target lesion length(s) ≤150 mm.
9. Target lesions(s) with reference vessel diameter (proximal and distal to target lesion) ≥2.0 mm and ≤4.0 mm.

Exclusion Criteria:

1. Subjects in whom amputation above the ankle is necessary, irrespective of the success of revascularization.
2. In-stent restenosis within the target lesion.
3. Flow-limiting dissection, Type C or greater.
4. Target lesions within an autogenous or prosthetic bypass graft.
5. History of an endovascular procedure or open vascular reconstruction in the index limb within the last 30 days, including thrombolytic therapy.
6. Any open vascular surgical procedure planned in the target limb or endovascular procedures planned in the target vessel within 30 days after the index procedure.
7. Kidney disease of sufficient severity, in the Investigator's opinion, to contraindicate lower extremity angiography using standard or alternate contrast agents as per the local Standard of Care.
8. Pregnancy or breast feeding. A woman of child-bearing potential must have a negative pregnancy test within one week of index procedure.
9. Myocardial infarction or stroke within 2 months of enrollment.
10. Contraindication to antiplatelet, anticoagulant, or thrombolytic therapy.
11. Uncorrectable bleeding diathesis, platelet dysfunction, thrombocytopenia with platelet count < 125,000/μL, known coagulopathy, or INR > 1.5.
12. Known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pretreated in the opinion of the investigator.
13. History of heparin-induced thrombocytopenia.
14. Psychiatric disorder which, according to the investigator, has potential to interfere with provision of informed consent, completion of tests, therapy, or follow-up.
15. Clinical/angiographic evidence of distal embolization or acute thrombus.
16. Significant stenosis (>50% diameter reduction) or occlusion of inflow vessels that was not successfully treated (<50% residual stenosis without flow limiting dissection) before the study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey G Carr, MD, Principal Investigator — Cardiovascular Associates of East Texas; Kenneth Ouriel, MD, Study Chair — Syntactx
Locations (17):
- United States (17):
  - Vascular Breakthroughs, Darien, Connecticut
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Precision Clinical Research, Lauderdale Lakes, Florida
  - Coastal Vascular and Interventional, Pensacola, Florida
  - St. Joseph's Hospital, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Community Health, Munster, Indiana
  - Michigan Outpatient Vascular Institute, Dearborn, Michigan
  - Vascular Access Center, Mays Landing, New Jersey
  - North Carolina Heart and Vascular, Raleigh, North Carolina
  - Allegheny Vein & Vascular, Bradford, Pennsylvania
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Pennsylvania Vascular Institute, Philadelphia, Pennsylvania
  - Anderson Heart, Anderson, South Carolina
  - DFW Vascular Group, Dallas, Texas
  - Houston Heart and Vascular, Kingwood, Texas
  - Cardiovascular Associates of East Texas, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carr J, Bowman J, Watts M, Ouriel K, Dave R. United States Investigational Device Exemption study of the Revolution Peripheral Atherectomy System. J Vasc Surg. 2022 Mar;75(3):976-986.e4. doi: 10.1016/j.jvs.2021.08.107. Epub 2021 Oct 5. PMID 34624496
- See also: RexMedical.com — http://www.rexmedical.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Revolution Treatment Arm
Started | 121
Completed | 121
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Revolution Treatment Arm
Number analyzed (Participants) | 121
Age, Customized [Mean (Standard Deviation); unit: Years]
  Age | 72 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 28
  White | 90
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 121

OUTCOME MEASURES:

1. Primary Outcome: Safety Endpoint: Number of Participants With Freedom From Major Adverse Events
Description: Freedom from Major Adverse Events is defined as the composite of all-cause mortality, clinically-driven target lesion revascularization (TLR), major target limb amputation, major target vessel perforation requiring surgical or endovascular repair, and clinically-significant distal embolization in the target limb; as adjudicated by an independent Clinical Events Committee The primary safety endpoint is freedom from 30-day Major Adverse Events (MAE), defined as the composite of all-cause mortality, clinically-driven target lesion revascularization (TLR), major target limb amputation, major target vessel perforation requiring surgical or endovascular repair and clinically-significant distal embolization in the target limb; as adjudicated by the independent Clinical Events Committee (CEC).
Time Frame: 30-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Revolution Treatment Arm
Number analyzed (Participants) | 113
Participants | 110

2. Primary Outcome: Effectiveness Endpoint: Technical Success
Description: Technical success is defined by ≤50% diameter stenosis after atherectomy with the Revolution™ Peripheral Atherectomy System and prior to adjunctive therapy, as measured by the independent core laboratory on the post-atherectomy contrast angiogram. Effectiveness will be assessed for investigator-identified target lesions and will be calculated as a binary variable as the percentage of target lesions with technical success.
Time Frame: 1-Day
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Revolution Treatment Arm
Number analyzed (Participants) | 121
Number analyzed (Lesions) | 123
Lesions | 111

3. Secondary Outcome: Target Lesion Revascularization (TLR) Rate
Description: Target Lesion Revascularization (TLR) rate through 30 days.
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Revolution Treatment Arm
Number analyzed (Participants) | 121
Participants | 0

4. Secondary Outcome: Change in % Stenosis
Description: Change in % stenosis after treatment with Revolution™ Peripheral Atherectomy System, determined after atherectomy and prior to other adjunctive therapies, as measured by the angiographic core laboratory.
Time Frame: 1-Day
Measure: Mean (Standard Deviation); unit: Percentage
Units Other Than Participants: Lesions
Arm/Group | Revolution Treatment Arm
Number analyzed (Participants) | 121
Number analyzed (Lesions) | 123
Percentage | 31.8 (19)

5. Secondary Outcome: Procedural Success
Description: Procedural success as defined by target lesion residual stenosis of <30% at the conclusion of the index procedure, after atherectomy and any adjunctive endovascular treatment, as measured by the angiographic core laboratory.
Time Frame: 1-Day
Population: 132 total lesions in the Per Protocol dataset. Images missing for 2 lesions; calibration missing for 3 lesions therefore only 127 post procedure angiograms available.
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Revolution Treatment Arm
Number analyzed (Participants) | 121
Number analyzed (Lesions) | 127
Lesions | 119

6. Secondary Outcome: Assessment of the Combined Components of the Primary Safety Endpoint, Freedom From MAE
Description: Assessment of the total combined components of the primary safety endpoint (Freedom from MAE); including all-cause mortality, major target limb amputation, clinically significant distal embolization, major target vessel perforation requiring surgical or endovascular repair, and clinically-driven TLR, measured through 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Revolution Treatment Arm
Number analyzed (Participants) | 121
Participants | 97

7. Secondary Outcome: Freedom From Target Lesion Revascularization (TLR) Rate
Description: Freedom from Target Lesion Revascularization (TLR) rate through 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Revolution Treatment Arm
Number analyzed (Participants) | 121
Participants | 105

8. Secondary Outcome: Freedom From Myocardial Infarction
Description: Freedom from Myocardial infarction through 30 days.
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Revolution Treatment Arm
Number analyzed (Participants) | 121
Participants | 121

9. Secondary Outcome: Freedom From Myocardial Infarction
Description: Freedom from Myocardial infarction through 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Revolution Treatment Arm
Number analyzed (Participants) | 121
Participants | 119

10. Secondary Outcome: Freedom From Target Vessel Revascularization (TVR) Rate
Description: Freedom from incidence of target vessel revascularization (TVR) through 30 days.
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Revolution Treatment Arm
Number analyzed (Participants) | 121
Participants | 121

11. Secondary Outcome: Freedom From Target Vessel Revascularization (TVR) Rate
Description: Freedom from incidence of target vessel revascularization (TVR) through 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Revolution Treatment Arm
Number analyzed (Participants) | 121
Participants | 121

12. Secondary Outcome: Freedom From Angiographic Procedural Distal Embolization
Description: Freedom from angiographic procedural distal embolization (symptomatic) in the target limb as confirmed angiographically by the core laboratory.
Time Frame: 1-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Revolution Treatment Arm
Number analyzed (Participants) | 121
Participants | 119

13. Secondary Outcome: Primary Patency
Description: Primary patency of the target lesion at 30 days and 6 months, determined by duplex ultrasound or angiography.
Time Frame: 30 Days, 6 months
Population: Among the 132 lesions in the Per Protocol dataset, four were excluded from the patency analyses due to missing post-atherectomy angiograms, leaving 128 lesions in the analysis.
Measure: Mean (Standard Error); unit: Percentage of primary patency
Units Other Than Participants: Lesions
Arm/Group | Revolution Treatment Arm
Number analyzed (Participants) | 121
Number analyzed (Lesions) | 128
Percentage of primary patency
  30 Days | 99.1 (0.9)
  6 Months | 81.6 (4.0)

14. Secondary Outcome: Assisted Primary Patency
Description: Primary-assisted patency of the target lesion at 30 days and 6 months, determined by duplex ultrasound or angiography.
Time Frame: 30 Days, 6 months
Population: as for outcome 13
Measure: Mean (Standard Error); unit: Percentage of assisted primary patency
Units Other Than Participants: Number of Per protocol lesions
Arm/Group | Revolution Treatment Arm
Number analyzed (Participants) | 121
Number analyzed (Number of Per protocol lesions) | 128
Percentage of assisted primary patency
  30 Days | 99.1 (0.9)
  6 Months | 87.7 (3.4)

15. Secondary Outcome: Secondary Patency
Description: Secondary patency of the target lesion at 30 days and 6 months, determined by duplex ultrasound or angiography.
Time Frame: 30 Days, 6 months
Population: as for outcome 13
Measure: Mean (Standard Error); unit: Percentage of secondary patency
Units Other Than Participants: Number of Per protocol lesions
Arm/Group | Revolution Treatment Arm
Number analyzed (Participants) | 121
Number analyzed (Number of Per protocol lesions) | 128
Percentage of secondary patency
  30 Days | 99.1 (0.9)
  6 Months | 91.6 (2.9)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Revolution Treatment Arm
All-Cause Mortality (participants affected / at risk) | 3/121
Serious Adverse Events (participants affected / at risk) | 26/121
Other Adverse Events (participants affected / at risk) | 78/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Revolution Treatment Arm (N=121)
Clinically Driven TLR (Vascular disorders) | 16
Major target limb amputation (Surgical and medical procedures) | 2
Perforation of target vessel (Vascular disorders) | 4
Distal embolization (Vascular disorders) | 1
All-cause mortality (General disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Revolution Treatment Arm (N=121)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 15
Cardiac disorders (Cardiac disorders) | 16
Endocrine disorders (Endocrine disorders) | 2
Eye disorders (Eye disorders) | 3
Gastrointestinal disorders (Gastrointestinal disorders) | 9
General disorders and administration site conditions (General disorders) | 23
Hepatobiliary disorders (Hepatobiliary disorders) | 1
Infections and infestations (Infections and infestations) | 16
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 14
Investigations (Investigations) | 2
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 3
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 8
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nervous system disorders (Nervous system disorders) | 4
Product issues (Product Issues) | 1
Psychiatric disorders (Psychiatric disorders) | 1
Renal and urinary disorders (Renal and urinary disorders) | 5
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 4
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 4
Surgical and medical procedures (Surgical and medical procedures) | 2
Vascular disorders (Vascular disorders) | 37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT02961894/Prot_002.pdf
  • Statistical Analysis Plan (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT02961894/SAP_003.pdf